CLINICAL TRIAL: NCT01372605
Title: SLAM DUNC: Strategies to Link Antidepressant and Antiretroviral Management at Duke University, University of Alabama at Birmingham, Northern Outreach Clinic (Henderson, NC), and University of North Carolina
Brief Title: Trial of Collaborative Depression Care Management for HIV Patients
Acronym: SLAM DUNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of North Carolina, Chapel Hill (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00019233; R01MH086362 (NIH)
Record Dates: First submitted 2011-06-12; First posted 2011-06-14 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Depression; HIV
Keywords: Depression; HIV; Adherence; Collaborative care; Measurement-Based Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collaborative depression care (Experimental): Measurement-Based Care: Decision support from paraprofessional to HIV medical provider around initiating and monitoring antidepressant treatment.
  Interventions: Other: Measurement-Based Care collaborative depression management
- Enhanced usual care (Other): Usual care. Enhanced through pre-study training of providers, provision of psychiatric diagnostic information at enrollment to HIV provider, and availability of best-practices guidelines for reference in clinic.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Other: Measurement-Based Care collaborative depression management — Depression Care Manager collects metrics on depressive severity and side effects and provides decision support regarding antidepressant initiation and modification to HIV providers who prescribe medications
  Arms: Collaborative depression care
Other: Enhanced Usual Care
  Arms: Enhanced usual care

SUMMARY:
This project will integrate a depression treatment and brief medication adherence counseling intervention into clinical care at three HIV clinics and will use a randomized controlled trial to assess whether, relative to usual care, the intervention leads to improved HIV medication adherence. The depression treatment intervention uses a model known as Measurement-Based Care which equips Depression Care Managers with systematic measurement tools, a decision algorithm, and psychiatric backup and trains them to provide decision support to HIV clinicians to implement, monitor, and adjust antidepressant therapy.

DETAILED DESCRIPTION:
Our goal in this project is to conduct a randomized controlled trial of an evidence-based depression treatment intervention known as Measurement-Based Care (MBC), combined with brief Motivational Interviewing (MI) adherence counseling, in depressed people living with HIV/AIDS to assess its impact on ART adherence and clinical outcomes. MBC employs Depression Care Managers with expertise in depression management to screen for depression and help non-psychiatric physicians implement guideline-concordant, algorithm-driven antidepressant treatment. The Depression Care Manager use standardized metrics (depressive symptoms, side effects) and an algorithm to monitor treatment response and recommend changes. Weekly supervision from a psychiatrist ensures quality care. Biweekly contact between patients and the Depression Care Manager will include brief MI adherence counseling.

We will recruit 390 people living with HIV/AIDS on antiretroviral therapy (ART) with confirmed depression, and will conduct a randomized trial of the MBC intervention versus enhanced usual care. Our aims are: (1) to test whether MBC improves ART adherence and HIV clinical outcomes, (2) to assess the cost-effectiveness of MBC, and (3) to collect process measures concerning MBC implementation to inform replication at other sites. Since the Depression Care Manager role can be effectively filled by a behavioral health provider or nurse given appropriate training and supervision and the intervention has limited time requirements, this model is potentially replicable to a wide range of resource-constrained HIV treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* HIV-positive
* Patient Health Questionnaire-9 (PHQ-9) total score >= 10
* Confirmed current major depressive episode
* English-speaking

Exclusion Criteria:

* History of bipolar disorder
* History of psychotic disorder
* Failure of adequate trials of two different antidepressants at effective doses in the current depressive episode
* Current substance dependence requiring inpatient hospitalization
* Not mentally competent
* Acute suicidality or other psychiatric presentation requiring immediate hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Pence, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Bradley N Gaynes, MD MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - University of Alabama at Birmingham 1917 Clinic, Birmingham, Alabama
  - University of North Carolina Hospitals Infectious Diseases Clinic, Chapel Hill, North Carolina
  - Duke University Clinic 2J, Durham, North Carolina
  - Northern Outreach Clinic, Henderson, North Carolina

REFERENCES:
- [Background] Pence BW, Gaynes BN, Williams Q, Modi R, Adams J, Quinlivan EB, Heine A, Thielman N, Mugavero MJ. Assessing the effect of Measurement-Based Care depression treatment on HIV medication adherence and health outcomes: rationale and design of the SLAM DUNC Study. Contemp Clin Trials. 2012 Jul;33(4):828-38. doi: 10.1016/j.cct.2012.04.002. Epub 2012 Apr 20. PMID 22542960
- [Background] Adams JL, Gaynes BN, McGuinness T, Modi R, Willig J, Pence BW. Treating depression within the HIV "medical home": a guided algorithm for antidepressant management by HIV clinicians. AIDS Patient Care STDS. 2012 Nov;26(11):647-54. doi: 10.1089/apc.2012.0113. PMID 23134559
- [Background] Bess KD, Adams J, Watt MH, O'Donnell JK, Gaynes BN, Thielman NM, Heine A, Zinski A, Raper JL, Pence BW. Providers' attitudes towards treating depression and self-reported depression treatment practices in HIV outpatient care. AIDS Patient Care STDS. 2013 Mar;27(3):171-80. doi: 10.1089/apc.2012.0406. Epub 2013 Feb 26. PMID 23442030
- [Background] Edwards M, Quinlivan EB, Bess K, Gaynes BN, Heine A, Zinski A, Modi R, Pence BW. Implementation of PHQ-9 depression screening for HIV-infected patients in a real-world setting. J Assoc Nurses AIDS Care. 2014 May-Jun;25(3):243-52. doi: 10.1016/j.jana.2013.05.004. Epub 2013 Oct 5. PMID 24103743
- [Background] Bengtson AM, Pence BW, O'Donnell J, Thielman N, Heine A, Zinski A, Modi R, McGuinness T, Gaynes B. Improvements in depression and changes in quality of life among HIV-infected adults. AIDS Care. 2015;27(1):47-53. doi: 10.1080/09540121.2014.946386. Epub 2014 Aug 8. PMID 25105320
- [Background] Pence BW, Quinlivan EB, Heine A, Edwards M, Thielman NM, Gaynes BN. When "need plus supply" does not equal demand: challenges in uptake of depression treatment in HIV clinical care. Psychiatr Serv. 2015 Mar 1;66(3):321-3. doi: 10.1176/appi.ps.201400132. Epub 2014 Dec 1. PMID 25727123
- See also: SLAM DUNC study website — http://slamdunc.web.unc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Started | 149 | 155
Completed | 137 | 145
Not Completed | 12 | 10
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Moved | 3 | 0
Not completed — Changed medical home | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Depression Care | Enhanced Usual Care | Total
Number analyzed (Participants) | 149 | 155 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.3) | 44.9 (9.9) | 43.9 (10.1)
Sex/Gender, Customized [Number; unit: participants]
  Male | 112 | 100 | 212
  Female | 35 | 52 | 87
  Transgender | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 140 | 151 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 86 | 107 | 193
  White | 58 | 43 | 101
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 149 | 155 | 304

OUTCOME MEASURES:

1. Primary Outcome: Antiretroviral Medication Adherence
Description: Antiretroviral medication adherence assessed by monthly unannounced pill count, assessed by blinded assessor
Time Frame: Six months post-enrollment
Population: All those completing a 6-month pill count which resulted in a valid adherence measure
Measure: Mean (Standard Deviation); unit: observed pills taken as % of expected
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 86 | 95
observed pills taken as % of expected | 89.2 (21.8) | 87.6 (22.9)

2. Secondary Outcome: Depressive Symptoms
Description: Hamilton Rating Scale for Depression (HAMD) symptom score at 6 months, assessed by blinded assessor. Possible score ranges from 0 to 50. Higher scores indicate worse depressive symptoms.
Time Frame: Six months
Population: All those completing a 6-month outcomes interview which resulted in a valid HAMD measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 92 | 98
units on a scale | 13.5 (7.6) | 17.2 (8.5)

3. Secondary Outcome: Antiretroviral Medication Adherence
Description: Antiretroviral medication adherence assessed by unannounced pill count, assessed by blinded assessor
Time Frame: 12 months
Population: Includes all individuals who completed a 6-month pill count that could be linked to an earlier (usually, 5-month) pill count, so as to calculate adherence. Some individuals did not complete this data point but still continued in the study and contributed later data.
Measure: Mean (Standard Deviation); unit: Percentage of expected pills
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 69 | 63
Percentage of expected pills | 86.3 (22.5) | 94.5 (12.4)

4. Secondary Outcome: Health Care Costs
Description: Total health care costs over 12 months
Time Frame: 12 months
Population: All participants were analyzed using all available time points, with multiple imputation used to address missing data.
Measure: Mean (Standard Error); unit: dollars
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 149 | 155
dollars | 4611 (151) | 4535 (148)

5. Secondary Outcome: Appointment Adherence
Description: Kept HIV appointments as a percentage of all kept or missed appointments during 12 months post-enrollment
Time Frame: 12 months
Population: All participants with available medical chart data on appointment attendance were analyzed. Some participants did not complete the study but still contributed chart abstraction data.
Measure: Mean (Standard Deviation); unit: Percent of appts that were kept
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 146 | 151
Percent of appts that were kept | 81.3 (23.9) | 80.1 (26.1)

6. Secondary Outcome: Number of Participants With Viral Load Below Detection
Description: HIV RNA viral load below the limit of detection at 6 months
Time Frame: 6 months
Population: All participants with a viral load available at 6 months. Some individuals without a viral load at 6 months still continued in the study and provided later data.
Measure: Number; unit: participants
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 79 | 98
participants | 68 | 75

7. Secondary Outcome: Quality of Life
Description: Short Form-12 Mental Composite score. Scores range from 0-100, with 50 corresponding to the mean and 10 points to the standard deviation in a normative US population. Higher scores indicate better health.
Time Frame: 6 months
Population: All participants who completed a 6-month research interview contributed data to this endpoint. Some participants did not complete the 6-month interview but still continued in the study and contributed later data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 92 | 98
units on a scale | 41.6 (12.4) | 37.6 (12.6)

8. Secondary Outcome: Self Reported Adherence
Description: Antiretroviral medication adherence, self-reported, over past 30 days using a visual analog scale. On the scale, participants report the percentage of prescribed antiretroviral pills that were taken in the past 30 days, ranging from 0 (no pills) to 100% (all pills).
Time Frame: 6 months
Population: All participants completing the 6-month interview and currently on antiretrovirals contributed to this analysis. Some participants did not complete the 6-month interview but still continued in the study and contributed to later data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 92 | 98
units on a scale | 92.7 (12.3) | 93.9 (15.0)

9. Secondary Outcome: Self-reported Adherence
Description: as for outcome 8
Time Frame: 12 months
Population: All participants completing the 12-month interview contributed data to this analysis. Some participants did not complete the 12-month interview but still completed the study and contributed other data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 69 | 81
units on a scale | 91.6 (16.4) | 94.1 (14.7)

10. Secondary Outcome: Safety Endpoint
Description: Psychiatric hospitalizations
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 149 | 155
participants | 2 | 4

11. Secondary Outcome: Depression-free Days
Description: Total depression-free days over 12 months as calculated from Hamilton Rating Scale for Depression scores at baseline and 3, 6, 9, and 12 months
Time Frame: 12 months
Population: All participants with at least one depression measure contributed to this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Number analyzed (Participants) | 143 | 137
days | 160 (9.9) | 136 (9.3)

ADVERSE EVENTS:
Description: Adverse events were collected without classification by specific Adverse Event Terms.
  Per protocol, hospitalizations were considered other adverse events in this study.
Arm/Group | Collaborative Depression Care | Enhanced Usual Care
Serious Adverse Events (participants affected / at risk) | 1/149 | 2/155
Other Adverse Events (participants affected / at risk) | 37/149 | 37/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Depression Care (N=149) | Enhanced Usual Care (N=155)
Death (Immune system disorders) | 1 (1) | 2 (2) — Death by all causes
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Depression Care (N=149) | Enhanced Usual Care (N=155)
Medical hospitalization (Immune system disorders) | 35 (63) | 33 (51) — This is hospitalizations from all non-psychiatric causes
Psychiatric hospitalization (Psychiatric disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No